CLINICAL TRIAL: NCT06703008
Title: "Monitoraggio Emodinamico Intraoperatorio in OLT"
Brief Title: Intraoperatory Hemodynamic Monitoring in OLT
Acronym: MEIO21
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MEIO21
Record Dates: First submitted 2023-08-30; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Liver Transplantation
Keywords: Hemodynamic Monitoring; TEE; Transesophageal Echocardiography; Transoesophageal Echocardiography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAC hemodynamic monitoring (No Intervention): Patients undergoing Liver Transplantation are monitored using the pulmonary artery catheter.
- TEE hemodynamic monitoring (Experimental): Patients undergoing Liver Transplantation are monitored using Transesophageal echocardiography and blinded to the pulmonary artery catheter data (insertion of PAC for patient safety is still mandatory, unblinding is allowed if needed for management by the OR anesthesiologist in charge)
  Interventions: Other: TEE hemodynamic monitoring

INTERVENTIONS:
Other: TEE hemodynamic monitoring — Transesophageal echocardiography monitoring to guide administration of fluids, vasopressor and inotropes during liver transplantation in order to avoid hypotension.
  Arms: TEE hemodynamic monitoring

SUMMARY:
The goal of this clinical trial is to compare two different hemodynamic monitoring techniques during orthotopic liver transplantation.

The main question it aims to answer is: if using a different hemodynamic monitoring might help reducing the intraoperative hypotension time. Participants will be randomized to one of two arms of hemodynamic monitoring:

* conventional monitoring with pulmonary artery catheter
* monitoring with transesophageal echocardiography Researchers will compare the two groups to see if there is any difference in the intraoperatory hypotension time and in secondary outcomes such as organ dysfunctions or mortality.

DETAILED DESCRIPTION:
Intraoperative hypotension is an independent risk factor for the development of complications and postoperative mortality. In non-cardiac surgery, in particular, the time spent under a mean arterial pressure (MAP) of 55 correlates with an increase in myocardial ischemic damage, acute renal failure, and 30-day mortality.

Orthotopic liver transplantation (OLT) is a complex and risky procedure both from a surgical and an anesthesiological standpoint. Difficulties in hemodynamic management arise from the pathophysiological alterations in cirrhotic patients, high-impact surgical procedures (e.g., caval and portal clamping), high bleeding risk, and post-reperfusion syndrome (PRS).

In liver transplantation, the pulmonary artery catheter (PAC) remains the "gold standard" for hemodynamic instability monitoring and is placed in over 90% of patients in the USA.

Transesophageal echocardiography (TEE) is a semi-invasive ultrasound monitoring procedure. As recognized in a recent position paper by the Society for the Advancement of Transplant Anesthesia (SATA), there has been a considerable increase in the use of TEE during OLT in recent years, despite the lack of randomized controlled trials (RCTs) confirming its effectiveness. According to the SATA task force, the increased intraoperative use of TEE is imputable to the chance for a more thorough understanding of hemodynamic pathophysiology and the possibility of identifying new findings, otherwise not identifiable with PAC (cardiac tamponade, gas embolism, intracardiac thrombus, papillary muscle/chordae rupture, left ventricular outflow tract obstruction, etc.). The overall complication rate of TEE in the articles analyzed by SATA was found to be 0.47% compared to 5-10% for PAC complications, thus supporting the safety of the procedure.

Currently, there is a lack of published RCTs comparing these monitoring methods to determine if there is an optimal intraoperative monitoring system during OLT.

The research hypothesis of this study is that TEE monitoring allows for better hemodynamic management during OLT, reducing the duration of hypotension and providing better guidance fo fluid-pharmacological therapy compared to standard monitoring (PAC).

The primary outcome is to compare the impact of two different hemodynamic monitoring systems (TEE and PAC) on intraoperative hemodynamic optimization during OLT.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for Liver Transplantation
* Acceptance of informed consent to participate in the study.

Exclusion Criteria:

* Bleeding esophageal varices
* Bleeding gastro-esophageal ulcer
* Gastro-esophageal anomalies (congenital, acquired or post-surgical)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of minutes with mean blood pressure (MAP) less than 65mmHg throughout surgery | From incision to end of procedure (for the entire surgical procedure in a period ranging from 0 to 24 hours).
  Cumulative time (in minutes) spent under mean arterial pressure of 65 mmHg.

SECONDARY OUTCOMES:
New Onset Renal Failure | From the end of the surgical procedure until discharge from hospital (whole duration of Hospital admission, considered within 3 months)
  New onset Renal Failure according to KDIGO( Kidney Disease Improving Global Outcomes) Criteria for Acute Renal Failure
New Onset Neurological disturbances | From the end of surgery for the first 24 hours after withdrawal of sedation in the ICU.
  Cumulative assessement of new-onset delirium, focal neurological disturbances or alteration of Glasgow Coma Scale GCS (from worst value GCS=3 to best value GCS=15 ) compared to the pre-operative status
New Onset Cardiological events | From the end of the surgical procedure until discharge from hospital (whole duration of Hospital admission, considered within 3 months)
  Cumulative outcome of : new onset acute coronary syndromes, ischemic alterations on post-operative EKG, new onset tricuspid insufficiency.
Cumulative Incidence of Early Graft Dysfunction / Primary Non Function | According to definition (up to 7 days after procedure).
  Cumulative Incidence of Early Graft Dysfunction / Primary Non Function as markers of graft failure.
Duration of Post-Reperfusion Syndrome | First 5 minutes after portal graft anastomosis.
  Duration of Post-Reperfusion Syndrome defined as hypotension (MAP< 65mmHg) lasting more than 1 minute in the first 5 minutes after portal graft anastomosis.
Total amount of fluids administered during surgery | From incision to end of procedure (for the entire surgical procedure in a period ranging from 0 to 24 hours)
  Total amount of crystalloids (in milliliters) administered during surgery
Cumulative dosage of vasoactive amines administered during surgery | From incision to end of procedure (for the entire surgical procedure in a period ranging from 0 to 24 hours)
  Total amount of norepinephrine and epinephrine (in mcg and in maximum dosage - mcg/kg/h - ) administered during surgery.
Cumulative incidence of adverse events attributable to the hemodynamic monitoring used | From the end of the surgical procedure until discharge from hospital (whole duration of Hospital admission, considered within 3 months)
  Cumulative incidence of adverse events attributable to the hemodynamic monitoring used
Duration of ICU admission | From a minimum of 2 days to a maximum of 3 months
  Duration of ICU admission in days
Mortality at 30 and 90 days | 1 month and 3 months after surgical procedure.
  Mortality at 30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Amedeo Bianchini, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCSS AOU di Bologna, Bologna, Emilia-Romagna, Italy